CLINICAL TRIAL: NCT05451498
Title: Effects of Creatine Monohydrate Timing on Resistance Training Adaptations in Male and Female Collegiate Athletes
Brief Title: Creatine Timing on Resistance Training Adaptations in College Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocky Mountain University of Health Professions (Other)
Collaborators: Lindenwood University (Other); Mayo Clinic (Other); Western Michigan University (Other)
Responsible Party: Principal Investigator, Nicholas Dinan, Principal Investigator, Rocky Mountain University of Health Professions
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol #2021-28
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: supplementation; pre-workout; post-workout; peri-workout; strength; endurance; body composition; fat-free mass
MeSH Terms: interventions — Creatine; maltodextrin

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel design
Who Masked: Participant, Investigator
Masking Description: A blinded research team that will not be involved in any other aspect of the study will be responsible for mixing and packaging the supplements for each participant. A blinded code will be established that represents all three supplement conditions and will be revealed after data has been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Creatine Pre-Exercise (Experimental): Consumes creatine within one hour before training and placebo within one hour after training
  Interventions: Dietary Supplement: Creatine
- Creatine Post-Exercise (Experimental): Consumes placebo within one hour before training and creatine within one hour after training
  Interventions: Dietary Supplement: Creatine
- Placebo (Placebo Comparator): Consumes placebo within one hour before training and placebo within one hour after training
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Creatine — Participants were matched according to fat-free mass to consume a placebo, or 5-g dose of creatine monohydrate within one hour before training, or within one hour after training for 8 weeks while completing a weekly resistance training program. At each time point (before and after training), all participants co-ingested a 25-gram dose whey isolate and a 25-gram dose of carbohydrate powder along with their assigned supplement. Body composition using a 3-compartment field (3CFIELD), muscular strength (one-repetition maximum [1RM]) and endurance (repetitions to fatigue [RTF] at 80% 1RM) using bench press (BP) and back squat (SQ) exercises along with isometric mid-thigh pull (IMTP) were assessed before and after the 8-week supplementation period.
  Arms: Creatine Post-Exercise; Creatine Pre-Exercise
Dietary Supplement: Maltodextrin — Participants were matched according to fat-free mass to consume a placebo (maltodextrin) within one hour before training, or within one hour after training for 8 weeks while completing a weekly resistance training program. At each time point (before and after training), all participants co-ingested a 25-gram dose whey isolate and a 25-gram dose of carbohydrate powder along with their assigned supplement. Body composition using a 3-compartment field (3CFIELD), muscular strength (one-repetition maximum [1RM]) and endurance (repetitions to fatigue [RTF] at 80% 1RM) using bench press (BP) and back squat (SQ) exercises along with isometric mid-thigh pull (IMTP) were assessed before and after the 8-week supplementation period.
  Arms: Placebo

SUMMARY:
While the use of creatine monohydrate supplementation and its associated benefits are well researched and supported, the impact of the timing of when creatine is ingested is a highly nuanced topic. The potential for the timing of administration to make an impact on observed outcomes is an established and appreciated factor and limited research to date has examined the impact of creatine timing. Of the literature that has been published, one study was very short in duration (4 weeks) that possessed a study design that undermined its practicality, two other studies used older individuals, and one study utilized a unilateral training model which may not be an adequate exercise protocol to allow for the ergogenic potential of creatine to mediate any enhancement of training adaptations. Therefore, based on the limited number of studies in young and previously trained populations, future studies examining the effects of pre vs post-training creatine monohydrate supplementation on resistance training adaptations are warranted.

DETAILED DESCRIPTION:
In a randomized, double-blind, placebo-controlled, parallel design, eligible study participants were provided a daily dose of creatine monohydrate (pre-or post-workout) or placebo (no creatine delivered) for an 8-week supplementation period. Based upon their baseline fat-free mass, participants were randomized into one of three groups: pre-workout creatine supplementation (PRE), post-workout creatine supplementation (POST), or placebo (PLA). Each group consumed their assigned dose or placebo within one hour before exercise and within one hour following exercise. Each assigned supplement was consumed with 12-16 ounces of fluid along with a 25-gram dose of whey protein isolate and a 25-gram dose of carbohydrate powder This additional supplementation was provided to aid in blinding and to help ensure adequate dietary protein intake was provided to promote increases in lean body mass and strength. Providing daily doses of carbohydrates and protein also helped with recruitment efforts as all study participants received some efficacious nutrients.

All participants completed a twelve-week resistance training and conditioning program. The first four weeks of resistance training (12 workouts) occurred before supplementation began and were completed to acclimate participants to the program and to initiate early neuromuscular adaptations commonly seen with starting a new resistance training program. In addition, this initial 4-week period allowed for some study participants to wash out from ongoing supplementation prior to beginning the supplementation protocol. After completion of this run-in period, participants then completed baseline testing as described and began the supplementation protocol while continuing to follow the resistance training program for an additional eight weeks. Before and after the 8-week supplementation and resistance training period, body mass, body water, and body composition were assessed in addition to changes in muscular strength, muscular endurance, and lower-body power. All statistical analysis was completed on data collected starting at the beginning and end of the supplementation period. Participants were provided nutritional recommendations in order to ensure adequate energy and protein consumption to facilitate positive training adaptations and reduce the potential influence of differing dietary intakes.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years of age but less than 30 years of age.
* Current member of Midland University athletic team completing off-season resistance training program.
* Participants will be healthy as determined by evaluation of medical history and if they are cleared to participate in their sport, they are cleared to participate in the study (as deemed by the team medical provider i.e. Certified Athletic Trainer).

Exclusion Criteria:

* As indicated on a medical history form they complete, any individual who is currently being treated or is diagnosed with a cardiac, respiratory, circulatory, musculoskeletal, metabolic obesity (defined as body mass index >35 kg/m2 and body fat greater than 30%), immune, autoimmune, psychiatric, hematological, neurological, or endocrinological disorder or disease will be excluded.
* Individuals with allergies to milk or soy (lecithin).
* For females only, if they are currently pregnant or become pregnant at any point throughout the study.

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Fat-Free Mass | 8 weeks
  3-compartment field (3CFIELD)
Lower Body Strength | 8 weeks
  Back Squat 1 repetition maximum according to standard protocols

SECONDARY OUTCOMES:
Fat Mass | 8 weeks
  3-compartment field (3CFIELD)
Body Fat Percentage | 8 weeks
  3-compartment field (3CFIELD)
Total Body Water | 8 weeks
  Determined by bioelectrical impedance spectroscopy
Upper Body Strength | 8 weeks
  Bench Press 1 repetition maximum according to standard protocols
Lower Body Muscular Endurance | 8 weeks
  80% 1 RM Back Squat repetitions to fatigue
Upper Body Muscular Endurance | 8 weeks
  80% 1 RM Bench press repetitions to fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas E Dinan, MS, Principal Investigator — Rocky Mountain University of Health Professions; Chad M Kerksick, PhD, Study Chair — Lindenwood University; Andrew R Jagim, PhD, Study Director — Mayo Clinic Health System; Michael G Miller, PhD, Study Director — Western Michigan University
Locations (1):
- Rocky Mountain University of Health Professions, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No